CLINICAL TRIAL: NCT04650022
Title: Predicting Value of DWI Total Posterior-circulation Infarct Volume for Endovascular Treatment Outcomes of Acute Basilar Artery Occlusion
Brief Title: Total Posterior-circulation Infarct Volume in Basilar Artery Stroke
Acronym: TPCIV-ABAO
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0636
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-11

CONDITIONS: Ischemic Stroke
Keywords: MRI; Posterior fossa; Thrombectomy; Stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TPCIV-ABAO: TPCIV-ABAO
  Interventions: Device: Mechanical thrombectomy

INTERVENTIONS:
Device: Mechanical thrombectomy — Stent retriever for treatment of cerebral arterial occlusions

SUMMARY:
Preprocedural predictors of outcome in patients with acute basilar artery occlusion (ABAO) who underwent endovascular treatment (EVT) remain controversial. The Investigators aimed to analyse, in patients with ABAO treated by EVT, if pre-EVT DWI total posterior-circulation infarct volume (TPIV) was a predictor of 90-days outcomes

DETAILED DESCRIPTION:
Acute basilar artery occlusion (ABAO) is a rare and devastating type of stroke. Endovascular treatment (EVT) is routinely performed in real-world practice, encouraged by the recent result of the basilar artery international cooperation study (BASICS), a randomized controlled study.

ABAO may result in infarcts in the brainstem, cerebellar lobes, thalamus and subthalamic area, or occipitotemporal lobes. Previously, studies using the DWI Posterior-circulation Alberta Stroke Program Early CT (Pc-ASPECT) Score or brainstem score, for predicting outcome in patients with ABAO, showed that the initial infarct extend can affect outcome. Some of these studies included patients tretaed by EVT. But, results showed conflicting findings.

To date, evidence regarding the association between pre-ETVT DWI lesion volume and outcomes is relatively weak and has not yet be determined. Predictors of the outcomes of EVT for anterior circulation include infarcts volume. More recently, authors reported a predictive model of good outcome combining initial DWI infarct volume of less than 10 ml, onset-to-puncture time less than 8 hours and embolic origin in 71 Korean patients undergoing EVT for vertebrobasilar occlusion. Nevertheless, up now, there is not sufficient evidence to reach a consensus.

Using data of our prospective registry, the investigators analyzed consecutive MRI selected, endovascularly treated ABAO patients within the first 24h after symptom-onset. Using the initial Magnetic Resonance Imaging (MRI), baseline total posterior-Circulation infarct volume (TPCIV) was calculated in mL, on an apparent diffusion-coefficient map reconstruction (Olea sphere software).

TPCIV was analyzed in univariate and multivariable models as a predictor of 90-day functional independence (modified Rankin Scale [mRS] 0-2) and mortality. According to received operating characteristic (ROC) analysis, the optimal cut-off was determined by maximizing the Youden index, to evaluate the prognostic value of TPCIV.

The Investigators aimed to investigate the relationship between baseline DWI total TPCIV and the 90-days functional outcome and mortality, in a large cohort of ABAO selected by MRI prior to EVT.

ELIGIBILITY:
Inclusion criteria:

* patient with a clinical diagnosis of acute stroke in the posterior-circulation within 24 hours from symptom onset;
* patient with a pertinent clinical deficit following physician evaluation (no NIHSS limit);
* acute basilar ischemia assessed on MRI matching clinical symptoms and including DWI;
* ABAO confirmed by intra-arterial arteriography and treated using mechanical thrombectomy.

Exclusion criteria:

Patients were excluded if they were ineligible for an MRI or ineligible for MT for the following reasons:

* prestroke modified Rankin Scale (mRS) score of >2;
* life expectancy <3 months;
* brainstem ischemia on DWI involving more than 80% of the area in axial view

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients >18 years, referred to our hospital, from January 2011 to October 2018, presenting acute basilar artery occlusion (ABAO) confirmed by magnetic resonance imaging treated by endovascular thrombectomy, with or without intravenous thrombolysis.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2011-01-30 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability | 90 day
  90-day functional outcome A favorable outcome was defined as a 90-day mRS≤2

SECONDARY OUTCOMES:
Mortality rate | 90 day
  Mortality and the cause of death at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Mourand, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC